CLINICAL TRIAL: NCT03376256
Title: Evaluation of the Compuflo Epidural Instrument for Thoracic Epidural Space Identification
Brief Title: Compuflo Instrument for Thoracic ES Identification
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in participant recruitment
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ralf E. Gebhard, MD, Professor of Clinical Anesthesiology, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170665
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia; Thoracic
Keywords: thoracic epidural; pressure measurement; device

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Phase A - Thoracic ES with LOR (Experimental): Patients will receive thoracic epidural anesthesia. The thoracic epidural needle will be introduced until loss of resistance (LOR) is perceived to identify the thoracic epidural space (ES). The Compuflo Epidural Instrument will be used to record pressure readings. The thoracic epidural procedure will then continue per standard of care.
  Interventions: Device: Compuflo Epidural Instrument
- Phase B - Thoracic ES with Compuflo (Experimental): Patients will receive thoracic epidural anesthesia. The thoracic epidural needle will be introduced until the Compuflo Epidural Instrument indicates that pressure has decreased. The loss of resistance technique will then be used to identify the thoracic epidural space. The thoracic epidural procedure will then continue per standard of care.
  Interventions: Device: Compuflo Epidural Instrument

INTERVENTIONS:
Device: Compuflo Epidural Instrument — Compuflo Epidural Instrument will be used to measure pressure levels in the thoracic epidural space while performing thoracic epidural anesthesia.

SUMMARY:
The purpose of this pilot study is to evaluate whether the Compuflo Epidural Instrument injection pump technology, which is FDA approved for lumbar epidural anesthesia, is also capable of identifying the thoracic epidural space through measurement of pressure levels. While this device is approved by the FDA for use in the procedure of the lumbar epidural, it is not used to perform the epidural procedure but rather to measure the epidural pressure. This study will likewise measure the epidural pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years inclusive
* BMI 18.5 to 40 inclusive
* Scheduled for thoracic epidural anesthesia

Exclusion Criteria:

* Patients younger than 18 years or older than 80 years of age
* Patients with BMI less than 18.5 or greater than 40
* Contraindication to thoracic epidural anesthesia
* Allergy or hypersensitivity to local anesthetics
* Patients with preexisting nerve damage
* Patients unable to provide written informed consent
* Individuals of vulnerable populations: children, pregnant women, prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf E Gebhard, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leurcharusmee P, Arnuntasupakul V, Chora De La Garza D, Vijitpavan A, Ah-Kye S, Saelao A, Tiyaprasertkul W, Finlayson RJ, Tran DQ. Reliability of Waveform Analysis as an Adjunct to Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):694-7. doi: 10.1097/AAP.0000000000000313. PMID 26469364
- [Background] Tsui BC, Gupta S, Finucane B. Confirmation of epidural catheter placement using nerve stimulation. Can J Anaesth. 1998 Jul;45(7):640-4. doi: 10.1007/BF03012093. PMID 9717595
- [Background] Kuo WC, Kao MC, Chang KY, Teng WN, Tsou MY, Chang Y, Ting CK. Fiber-needle swept-source optical coherence tomography system for the identification of the epidural space in piglets. Anesthesiology. 2015 Mar;122(3):585-94. doi: 10.1097/ALN.0000000000000531. PMID 25437497
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Lechner TJ, van Wijk MG, Maas AJ. Clinical results with a new acoustic device to identify the epidural space. Anaesthesia. 2002 Aug;57(8):768-72. doi: 10.1046/j.1365-2044.2002.02621.x. PMID 12133089
- [Background] Crawford JS. The second thousand epidural blocks in an obstetric hospital practice. Br J Anaesth. 1972 Dec;44(12):1277-87. doi: 10.1093/bja/44.12.1277. No abstract available. PMID 4265424
- [Background] Thangamuthu A, Russell IF, Purva M. Epidural failure rate using a standardised definition. Int J Obstet Anesth. 2013 Nov;22(4):310-5. doi: 10.1016/j.ijoa.2013.04.013. Epub 2013 Aug 6. PMID 23932551
- [Background] Ready LB. Acute pain: lessons learned from 25,000 patients. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):499-505. doi: 10.1016/s1098-7339(99)90038-x. No abstract available. PMID 10588551

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase A - Thoracic ES With LOR | Phase B - Thoracic ES With Compuflo
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in phase B prior to study termination
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase A - Thoracic ES With LOR | Phase B - Thoracic ES With Compuflo | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pressure Levels in Thoracic Epidural Space
Description: The Compuflo Epidural Instrument measures the pressure levels in millimeters of mercury (mmHg) in the thoracic epidural space
Time Frame: Day 1
Population: No participants were enrolled in phase B prior to study termination
Measure: Number; unit: mmHg
Arm/Group | Phase A - Thoracic ES With LOR | Phase B - Thoracic ES With Compuflo
Number analyzed (Participants) | 2 | 0
mmHg | NA — Results not reported due to participant confidentiality |

2. Secondary Outcome: Percent of Successful Performance of Thoracic Epidural Anesthesia Using Loss of Resistance Technique
Description: Percent of thoracic epidural anesthesia procedures using LOR that result in a loss of sensation to cold in at least one dermatome, either unilateral or bilateral
Time Frame: Day 1
Population: No participants were enrolled in phase B prior to study termination
Measure: Number; unit: Percent of successful performance
Arm/Group | Phase A - Thoracic ES With LOR | Phase B - Thoracic ES With Compuflo
Number analyzed (Participants) | 2 | 0
Percent of successful performance | NA — Results not reported due to participant confidentiality |

ADVERSE EVENTS:
Time Frame: 2 days
Description: Adverse events not reported due to participant confidentiality
Arm/Group | Phase A - Thoracic ES With LOR | Phase B - Thoracic ES With Compuflo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
To protect participant privacy and maintain confidentiality, results will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03376256/Prot_SAP_000.pdf